CLINICAL TRIAL: NCT03526887
Title: A Phase II Open-label Multicenter Exploratory Study to Assess Efficacy of Pembrolizumab Re-challenge as Second or Further Line in Patients With Advanced Non - Small Cell Lung Cancer
Brief Title: Re-challenge Pembrolizumab Study as a Second or Further Line in Patients With Advanced NSCLC
Acronym: Replay
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP 17/02_REPLAY; 2017-003947-39 (EudraCT Number)
Record Dates: First submitted 2018-04-17; First posted 2018-05-16 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 2 groups depending on when the progression disease is diagnosed but the treatment after progression will be the same: Pembrolizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients who experienced progression disease while on treatment progression disease < 12 weeks after stopping treatment. After that the patients took chemotherapy ≥ 4 cycles and progressed again. After the last progression the patient is included in the study to be retreated with Pembrolizumab 200mg
  Interventions: Drug: Pembrolizumab
- Cohort 2 (Experimental): Stop treatment and progression > 12 weeks after stopping treatment. After the last progression the patient is included in the study to be retreated with Pembrolizumab 200mg
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg, Q3W
  Other Names: KEYTRUDA
  Arms: Cohort 1
Drug: Pembrolizumab — 200 mg, Q3W
  Other Names: KEYTRUDA
  Arms: Cohort 2

SUMMARY:
Exploratory phase II trial of intravenous (IV) Pembrolizumab MK-3475 as second or further line with advanced Non-small cell Lung Cancer (NSCLC) who have failed to a prior treatment with anti-PDL1 drug.

Pembrolizumab 200 mg ,Q3W, IV infusion, Day 1 of each 3 week cycle will be administered until disease progression.

DETAILED DESCRIPTION:
This is a multi-center exploratory phase II trial of intravenous (IV) Pembrolizumab MK-3475 as second or further line with advanced Non-small cell Lung Cancer (NSCLC) who have failed to a prior treatment with anti-PDL1 drug.

110 patients will be enrolled in this trial to examine the efficacy and outcomes of these patients.

In addition to the usual procedures in a phase II study (evaluation of response, toxicity, etc.) special attention will be paid in this trial to the molecular assessment in biological samples.

Subjects will receive Pembrolizumab at a fixed dose of 200 mg every 3 weeks (Q3W). Subjects will be evaluated with radiographic imaging to assess response to treatment. Investigators will make all treatment-based decisions using the Immune-Related Response Criteria (irRC). However, for determination of overall response rate (ORR) and progression-free survival (PFS), the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 will be used.

Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Treatment with Pembrolizumab will continue until documented disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, noncompliance with trial treatment or procedure requirements, or administrative reasons.

After the end of treatment, each subject will be followed for a minimum of 30 days for adverse event monitoring (serious adverse events will be collected for up to 90 days after the end of treatment unless the subject starts a new anticancer therapy between days 31 and 90). Subjects will have post-treatment follow-up for disease status, including initiating a non-study cancer treatment and experiencing disease progression, until death, withdrawing consent, or becoming lost to follow-up.

Participation in this trial will be dependent upon supplying tumor tissue from a newly obtained formalin-fixed specimen from locations not radiated prior to biopsy. The specimen will be evaluated at a central laboratory facility for expression status of PD-L1 in a prospective manner. Only subjects whose tumors express PD-L1 as determined by the central laboratory facility will be eligible for inclusion in this study. Also it is highly recommend to send archival tumor tissue from the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cythological confirmed NSCLC advanced or locally advanced disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) not amenable to radical treatment (IIIA, IIIB, IIIC, IV), squamous or non-squamous, recurrent after at least one prior line.
2. The subject must be willing and able to provide written informed consent/assent for the trial.
3. Patient must be aged ≥ 18 years of age on day of signing informed consent.
4. Measurable disease (at least 1 lesion) based on RECIST 1.1. Patients will not be eligible if this lesion was irradiated before inclusion.
5. Documented prior benefit (Stable Disease, Partial Response, Complete Response) to check point PD1/PDL1 inhibitor (Nivolumab, Pembrolizumab, Durvalumab, Atezolizumab, Avelumab or others) for at least 16 weeks (Stable Disease, Partial Response, Complete Response) and progression while on treatment (or <12 weeks after stopping) with the same PD-1/PD-L1 inhibitors. These patients should have received subsequent treatment with Chemotherapy for at least 4 courses (Cohort 1) OR Documented prior benefit (Stable Disease, Partial Response, Complete Response) to check point PD1/PDL1 inhibitor (Nivolumab, Pembrolizumab, Durvalumab, Atezolizumab, Avelumab or others) for at least 16 weeks (Stable Disease, Partial Response, Complete Response) and progression >12 weeks after stopping treatment (Cohort 2). No subsequent treatment before rechallenge is allowed in this cohort
6. Patient must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. PDL1 must be evaluable and at least 1% positive in tumor tissue. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor. Note: If a new sample core or excisional biopsy cannot be obtained but the patient can be included in the study and start the treatment and the archival tumor tissue could be sent afterwards for the central laboratory confirmation. If no previous PDL1 result is available from the archival tissue, the patient cannot be included in the trial until central laboratory PDL1 result is available. Other cases could be consulted with the trail chair.
7. Have a performance status of 0-1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function, all screening labs should be performed within 7 days of treatment initiation.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential must be willing to use an adequate method of contraception (for the course of the study through 120 days after the last dose of study medication).

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential must agree to use an adequate method of contraception (starting with the first dose of study therapy through 120 days after the last dose of study therapy).

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. All patients will be required to submit a tumor sample for PD-L1 IHC expression. If the sample is inadequate for analysis, another sample could be provided. If a new sample cannot be obtained due to technical or clinical reasons, archival tissue can be sent. Other cases could be consulted with the trial chair.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids at a dose over 10 mg of prednisone or equivalent, for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Documented EGFR sensitizing mutation.
13. Documented ALK translocation.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
20. Received radiation therapy to the lung of >30Gy within 6 months of the first dose of trial treatment.
21. Evidence of interstitial lung disease.
22. Has had previously serious adverse reactions (grade 3-4) related to previous PD1/PDL1 inhibitors that preclude their treatment according to the principal investigator' s criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luís Paz Ares, MD, Principal Investigator — Hospital 12 de Octubre
Locations (19):
- Spain (19):
  - Hospital General Universitario de Elche, Elche, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Complejo Hospitalario de la Coruña, A Coruña, Coruña
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital de Santa Creu i Sant Pau, Barcelona
  - H.U.Vall D´Hebrón, Barcelona
  - Hospital Dr. Josep Trueta, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Fundación Jiménez Díaz, Madrid
  - H. 12 de Octubre, Madrid
  - Puerta de Hierro, Madrid
  - H. Son Llàtzer, Palma de Mallorca
  - Hospital General Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — https://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 55 | 18
Completed | 55 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 55 | 18 | 73
Age, Continuous [Median (Full Range); unit: years] | 63.5 [41 to 80] | 69.8 [55 to 83] | 65 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 15 | 54
  Male | 16 | 3 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 53 | 18 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Spain | 55 | 18 | 73
Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  Participants
    ECOG 0 | 15 | 8 | 23
    ECOG 1 | 39 | 10 | 49
    ECOG 2 | 0 | 0 | 0
    ECOG 3 | 0 | 0 | 0
    ECOG4 | 0 | 0 | 0
    Not recorded | 1 | 0 | 1
Cigarette Smoking History [Count of Participants; unit: Participants]
  Never smoker | 7 | 1 | 8
  Former smoker | 39 | 15 | 54
  Smoker | 8 | 2 | 10
  Not recorded | 1 | 0 | 1
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26 [17.1 to 35.3] | 28 [20.2 to 34.8] | 26.5 [17.1 to 35.3]
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 32 | 8 | 40
  Squamous | 19 | 8 | 27
  Adeno-squamous | 2 | 0 | 2
  Large Cell Carcinoma | 1 | 1 | 2
  NOS/Undifferentiated | 1 | 0 | 1
  Other | 0 | 1 | 1
Clinical Stage [Count of Participants; unit: Participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body.
  There are 5 stages for NSCLC:
  Stage 0:tumor hasn't grown into nearby normal lung tissues Stage I:small tumor that hasn't spread to any lymph nodes Stage II: medium tumor that hasn't spread to the nearby lymph nodes or N1 Stage III: cancer spread to the lymph nodes but haven't spread to other distant parts of the body Stage IV: cancer has spread to more than 1 area in the other lung, the fluid surrounding the lung or the heart or distant parts of the body
  Participants
    Stage I | 0 | 0 | 0
    Stage II | 0 | 0 | 0
    Stage III | 3 | 1 | 4
    Stage IV | 52 | 17 | 69

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pembrolizumab Re-challenge Measured by Overall Survival
Description: Overall survival: Defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 55 | 18
months | 9.4 [1 to 18] | 19.1 [3 to 48]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.016, Log Rank; Median Difference (Net) = 9.7, 95% CI 2-sided [9.4 to 19.1]

2. Secondary Outcome: Efficacy of Pembrolizumab Re-challenge Measured by Progression Free Survival (PFS) Per RECIST v1.1.
Description: PFS: Defined as the length of time from the date of randomization to the date of the first documented progression of disease. "Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions"
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 55 | 18
months | 1.6 [0 to 11] | 4.1 [0.2 to 18]

3. Secondary Outcome: Best Global Response
Description: To evaluate the best global response of the treatment as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of randomization until end of follow up, up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 55 | 18
Participants
  Complete response | 0 | 0
  Partial response | 1 | 3
  Stable disease | 24 | 11
  Progression disease | 25 | 3
  Not evaluable | 5 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed an average of 30 months. Deaths were assessed up to 48 months.
Description: Any adverse event or breakdown occurring during the course of the study. The investigator will have to collect all adverse events once they have signed informed consent, during treatment and 30 days after the last dose study treatment administration.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 44/55 | 5/18
Serious Adverse Events (participants affected / at risk) | 2/55 | 1/18
Other Adverse Events (participants affected / at risk) | 29/55 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=55) | Cohort 2 (N=18)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=55) | Cohort 2 (N=18)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 7 (7) | 4 (4)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03526887/Prot_SAP_000.pdf